CLINICAL TRIAL: NCT05938894
Title: The Effect of Executive Function Training on Diet and Attitudes
Brief Title: Train Your Brain - Executive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC299
Record Dates: First submitted 2023-05-07; First posted 2023-07-11 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Overweight and Obesity
Keywords: Normal weight
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFfect-food choices (Experimental): Participants will complete four online games at least biweekly during the study.
  Interventions: Other: online games with various food images
- Control (Active Comparator): Participants will complete four online games at least biweekly during the study.
  Interventions: Other: online games with images of flowers and songbirds

INTERVENTIONS:
Other: online games with various food images — Participant will play a series of online games with various food images.
  Arms: EFfect-food choices
Other: online games with images of flowers and songbirds — Participant will play a series of online games with images of flowers and songbirds.
  Arms: Control

SUMMARY:
The purpose of this research is to test if playing games designed to improve an individual's executive function can change their views about the types of foods they eat. Executive function is a set of mental processes that people use every day to make decisions - such as what kinds of foods they choose to eat and when and where they eat those foods.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether executive function (EF) training concurrently improves attitudes, perceptions, and consumption of nutrient-dense foods (i.e., fruits, vegetables) while worsening the same of nutrient-poor foods. In effect, the aim is to test whether EF training can promote the substitution of nutrient-poor foods with fruits and vegetables (FV), as the Dietary Guidelines for Americans (DGA) recommends regular consumption of FV as part of a healthy dietary pattern. Given the health benefits associated with consuming FV, EF training that effectively promotes increased FV intake may benefit health. For example, FV consumption is associated with the reduced risk of all-cause mortality, cardiovascular disease, diabetes, cancer, and eye and skin health. Moreover, FV consumption is associated with better mental and cognitive health.

ELIGIBILITY:
Inclusion Criteria:

* BMI 23-38 kg/m2
* US citizenship
* Not currently dieting to lose weight and no weight loss or gain of >2 kg over the past 3 months
* No tobacco or e-cigarette use
* Not pregnant or lactating or planning to become pregnant while participating in the study

Exclusion Criteria:

* Not a US citizen
* Currently dieting to lose weight
* Weight loss of >2 kg over the past 3 months
* Tobacco or e-cigarette use
* Pregnant or lactating or planning to become pregnant while participating in the study
* A history of bariatric surgery
* Diagnosis of major medical or psychiatric condition that would interfere with participation, including not being physically able to play the games, or a current eating disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Change in response time | Week 0, Week 9
  Change in online game speed of response time
Change in percent correct | Week 0, Week 9
  Change in online game percent correct

CONTACTS AND LOCATIONS:
Overall Officials: Shanon Casperson, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roemmich JN, Nelson AM, Stice E, Hess JM, Palmer DG, Casperson SL. Efficacy of a Web-Based Executive Function Training Program to Induce Healthier Food Choices and Increase Valuation of Fruits and Vegetables in Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 16;14:e66394. doi: 10.2196/66394. PMID 40957017
- See also: Grand Forks Human Nutrition Research Center Train Your Brain Study website — https://trainyourbrain.usda.gov/
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT05938894/ICF_000.pdf